CLINICAL TRIAL: NCT02244528
Title: Pharmacokinetic Study of Sildenafil in Neonates and Preterm Infants
Brief Title: PK Study of Sildenafil in Neonate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14172MFDS178-1
Record Dates: First submitted 2014-09-11; First posted 2014-09-19 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Neonates and Preterm Infants
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): sildenafil treatment
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of sildenafil which is used as treatment of pulmonary hypertension in neonate and preterm infant.

ELIGIBILITY:
Inclusion Criteria:

* Admitted at NICU in Seoul National University Hospital or Bundang Seoul National University hospital
* Infants who were diagnosed with PAH

Exclusion Criteria:

* Severe allergic reaction to sildenafil
* Inotropics for hypotension within 3 days prior to enrollment
* AST or ALT > 3x ULN
* Any condition that would make the participant, in the opinion of the investigator, unsuitable for the stud

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | t up to 5 weeks
  5 times drug level after 5 doses (pre30min/post 30min, 1hr, 2hr, 4hr) pharmacokinetics
Cmax(0-t) | t up to 5 weeks
  5 times drug level after 5 doses (pre30min/post 30min, 1hr, 2hr, 4hr) pharmacokinetics

SECONDARY OUTCOMES:
Change from baseline in pulmonary arterial hypertension at 5 weeks | pre, 2 weeks, 5 weeks of drug administration
  Echocardiography
  * RV systolic pressure: TR velocity2 x 4
  * Septum contour: normal, flat at end-systole, flat at end-diastole
  * LV shape: normal, partially D-shape, D-shape, squeezed
  * LV eccentricity index
  * RV area/LV area (Apical 4 chamber view, at end diastole)
  * RA enlargement (Apical 4 chamber view)
  * RV anterior wall thickness
  * TAPSE (Tricuspid annular plane systolic excursion)
  * RV Tei index (by tissue Doppler)
  * Tissue Doppler velocity at RV free wall
respiratory severity score | pre, 2 weeks, 5 weeks after administration
  Mean airway pressure x FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Children's Hospital, Seoul